CLINICAL TRIAL: NCT02179541
Title: RGB Measurements as a Novel Objective Diagnostic Test for Otitis Media With Effusion
Brief Title: A Novel Objective Diagnostic Test for Otitis Media With Effusion
Status: Completed | Type: Observational
Sponsor: Nazan Degirmenci (Other)
Responsible Party: Sponsor-Investigator, Nazan Degirmenci, M.D, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Other Study IDs: B.30.2.BAV.0.05.05/467; B.30.2.BAV.0.05.05/467 (Other: Bezmialem Vakif University)
Record Dates: First submitted 2014-05-30; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2013-01

CONDITIONS: Otitis Media With Effusion
Keywords: Otitis media with effusion, viscosity, RGB (red-green-blue).
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: All Group 1 patients were diagnosed with OME, diagnoses made by endoscopic-otoscopic examination findings and type-B tympanograms. They were all scheduled for ventilation tube insertion. Diagnosis of OME was confirmed during this surgery. All patients were examined by 4 mm 0-degree Storz endoscope and light source. The Adobe Photoshop Elements 7.0 program was used for RGB measurements. Viscosity was measured by the Brookfield DV-II+ProCP Viscometer.
  Interventions: Other: RGB
- Group 2: Children in Group 2 had totally normal tympanic membranes and type A tympanograms. They had no hearing loss, Eustachian tube dysfunction, or any other ear-related problem, and were included in the study as healthy controls. Excluded from the study were patients presenting with acute otitis media, tympanosclerotic plaques, mental retardation, and children who were difficult to cooperate with. All subjects were examined by 4 mm 0-degree Storz endoscope and light source. The Adobe Photoshop Elements 7.0 program was used for RGB measurements.
  Interventions: Other: RGB
- Group 1a: To determine whether higher or lower viscosity of an effusion impacted RGB values, the patient group was subdivided into two subgroups according to viscosity level. Patients with an effusion below the mean viscosity value of 450 cP (centipoise) were assigned to Group 1a.
  Interventions: Other: RGB
- Group 1b: To determine whether higher or lower viscosity of an effusion impacted RGB values, the patient group was subdivided into two subgroups according to viscosity level. Patients with an effusion above the mean viscosity value of 450 cP (centipoise) were assigned to Group 1b.
  Interventions: Other: RGB

INTERVENTIONS:
Other: RGB — When a circular area of 30 surrounding pixels are placed exactly upon the above-mentioned standardized points, the Adobe Photoshop Elements 7.0 program automatically measures the numerical values of the RGB color components in that area. The RGB values of the same points on the tympanic membrane images of the two groups were obtained and compared. Diagnostic significance of objectively assessed color changes at the tympanic membrane in OME patients was evaluated.

SUMMARY:
Otitis media with effusion (OME) cases refer to a clinically silent condition. Otoscopic findings are subjective and not always reliable. As an objective test tympanometric evaluation is imperfect for diagnosis of OME. The objective of our study was to investigate, in OME cases, the correlation of tympanic membrane color changes with the presence and viscosity of effusion in the middle ear. The study aimed to provide objective diagnostic and therapeutic criteria for patients scheduled for surgery by 2 means: measuring the viscosity of the fluid and evaluating color changes objectively with red-green-blue (RGB) measurements.

DETAILED DESCRIPTION:
Endoscopic images of the tympanic membranes of 52 patients (Group 1) and 52 healthy controls (Group 2) were taken during their otologic examinations. All patients in Group 1 had hearing loss and were diagnosed with OME after audiological evaluation. Specific points were designated at certain areas on each tympanic membrane, and RGB values of those specific points were measured on the tympanic membrane images of both groups. Additionally, in Group 1 viscosity of each effusion taken by paracentesis during surgery was also measured intraoperatively with a viscometer. Patients with viscosity values lower than 450 cP (centipoise) were subdivided into Group 1a, and those with values higher than 450 cP into Group 1b.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OME, that had endoscopic-otoscopic examination findings and type-B tympanograms.
* They were all scheduled for ventilation tube insertion.

Exclusion Criteria:

* Patients presenting with acute otitis media, tympanosclerotic plaques, mental retardation, and children who were difficult to cooperate with.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Endoscopic images of the tympanic membranes of 52 patients (Group 1) and 52 healthy controls (Group 2) were taken during their otologic examinations. RGB values of specific points were measured on the tympanic membrane images of both groups. Additionally, in Group 1 viscosity of each effusion taken by paracentesis during surgery was also measured intraoperatively with a viscometer. Patients with viscosity values lower than 450 cP (centipoise) were subdivided into Group 1a, and those with values higher than 450 cP into Group 1b.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean RGB values | January-May 2013 (5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Selahattin TUGRUL, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)